CLINICAL TRIAL: NCT00543829
Title: A Randomised, Controlled, Open Phase II b Study Comparing a Combination of Dose-Intensified Doxorubicin and Docetaxel With or Without Tamoxifen as Preoperative Therapy in Patients With Operable Carcinoma of the Breast (T>=3cm N0-2 M0)
Brief Title: German Preoperative Adriamycin Docetaxel Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gepardo
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; doxorubicin; docetaxel; tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Docetaxel; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 4 cycles of doxorubicin and docetaxel with tamoxifen
  Interventions: Drug: doxorubicin, docetaxel, tamoxifen
- 2 (Active Comparator): 4 cycles of doxorubicin and docetaxel without tamoxifen
  Interventions: Drug: doxorubicin, docetaxel

INTERVENTIONS:
Drug: doxorubicin, docetaxel, tamoxifen — Every 14 days to a total of 4 cycles of doxorubicin (50 mg/m², 15 minutes i.v. infusion) and docetaxel (75 mg/m², 1 hour i.v. infusion) with tamoxifen (30 mg tablet p.o. for 5 years post surgery)
  Arms: 1
Drug: doxorubicin, docetaxel — Every 14 days to a total of 4 cycles of doxorubicin (50 mg/m², 15 minutes i.v. infusion) and docetaxel (75 mg/m², 1 hour i.v. infusion)
  Arms: 2

SUMMARY:
The primary objective of this trial is to determine the rate of pathologically complete remissions following a preoperative dose-intensified therapy with doxorubicin and docetaxel with or without tamoxifen in patients with operable carcinoma of the breast. Secondary aims are to assess the rate of clinical complete and partial responses, of breast-conserving operations, and the toxicity of chemotherapy with and without tamoxifen.

Women meeting the following criteria will be eligible for the study: operable breast cancer (T³3cm N0-2 M0), histologically confirmed diagnosis by core-cut needle or incisional biopsy, and measurable disease by mammography or sonography or breast MRI (best appropriate method has to chosen by investigator). After the patients have given written informed consent, they will be randomised to the study treatments. All patients are scheduled to receive 4 cycles of combination chemotherapy consisting of doxorubicin 50 mg/m² (15-min i.v. infusion) and docetaxel 75 mg/m² (1-h i.v. infusion). The patients allocated to group I additionally receive oral doses of tamoxifen 30 mg once daily, starting on the first day of chemotherapy, while chemotherapy alone is administered to patients of group II. Cycles should be repeated every 14 days, followed by surgery 8 weeks after initiation of the trial. Surgery consists of removal of the remaining tumour (breastconserving resection or mastectomy) and axillary dissection. Patients with no response or even progression of the primary tumour can be treated to the discretion of the investigator but should be followed up according to protocol. If a partial or complete tumour response has been achieved, radiotherapy is given to the remaining breast in patients undergoing breast conserving therapy, and tamoxifen treatment is continued for a further 5 years.

Response will be assessed between the 4th cycle and surgery, using the best appropriate method. Clinical evaluation should be performed after each cycle. It is planned to recruite 200 patients during a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary carcinoma of the breast, confirmed histologically by core-cut needle or incisional biopsy. Fine needle aspiration is not sufficient.
* Bidimensionally measurable tumour, either by mammography or breast ultrasound or breast MRI
* Primary tumour >= 3 cm in largest diameter. In patients with multifocal or multicentric breast cancer the largest lesion should be measured.
* No evidence of distant metastases (as confirmed by chest x-ray, liver ultrasound and bone scintigraphy)
* Age >= 18 years and <= 70 years.
* Life expectancy at least 10 years, ignoring the diagnosis of cancer.
* Karnofsky index >=70%.
* Adequate haematologic, renal and hepatic function (WBC >4000, platelets >100000, bilirubin, serum creatinine and transaminases within the normal range).
* Anamnestic and electrocardiographic evidence of normal cardiac function, without or with medication. Normal cardiac function measured by echocardiography or MUGA-scan.
* Negative pregnancy test and appropriate non-hormonal contraception in fertile women.
* Written informed consent and presumed compliance of the patients.

Exclusion Criteria:

* Locally advanced (stage T4), bilateral, metastatic, or inflammatory breast cancer (tethering or dimpling of the skin as well as nipple inversion may not easily be interpreted as skin infiltration). If one of these conditions is suspected it has to be excluded before enrollment onto study.
* Previous treatment for breast cancer, including surgery, radiation, cytotoxic or endocrine treatments. Surgical diagnostic procedures are allowed.
* Previous malignancy other than breast cancer or non-invasive breast lesions if the disease-free interval is less than 10 years.
* Previous cytotoxic treatment for any condition.
* Preexisting neurotoxicity greater than grade II (WHO).
* Active infection or other significant illness that could influence tolerability of treatment.
* Current treatment with sex hormones (treatment has to be discontinued before the start of systemic therapy).
* Psychiatric illness or drug addiction that would preclude obtaining informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 1998-04; Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is defined as no microscopic evidence of viable tumour in the resected breast specimen | Post surgery

SECONDARY OUTCOMES:
Endpoints are (1) clinical partial or complete response and (2) clinical complete response | Post surgery
Endpoint is breast conservation without the need for autologous or heterologous reconstruction | Post surgery
Endpoints are the frequency of grade III and IV haematological and non-haematological toxicities during chemotherapy and delayed cardiotoxicity | 2 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Kaufmann, MD, Principal Investigator — J. W. Goethe University, School of Medicine, Dep. of Gynecology and Obstetrics

REFERENCES:
- [Derived] von Minckwitz G, Sinn HP, Raab G, Loibl S, Blohmer JU, Eidtmann H, Hilfrich J, Merkle E, Jackisch C, Costa SD, Caputo A, Kaufmann M; German Breast Group. Clinical response after two cycles compared to HER2, Ki-67, p53, and bcl-2 in independently predicting a pathological complete response after preoperative chemotherapy in patients with operable carcinoma of the breast. Breast Cancer Res. 2008;10(2):R30. doi: 10.1186/bcr1989. Epub 2008 Apr 1. PMID 18380893